CLINICAL TRIAL: NCT06291857
Title: A Randomized, Observer-Blinded, Active-Controlled Study to Evaluate the Safety and Immunogenicity of a COVID-19 Influenza Combination Nanoparticle Vaccine and a Standalone Trivalent Nanoparticle Influenza Hemagglutinin Vaccine in Participants ≥ 65 Years of Age.
Brief Title: A Study to Evaluate the Safety and Immunogenicity of COVID-19 Vaccine and Influenza Combination Vaccine
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novavax (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: CIC-E-301
Record Dates: First submitted 2024-03-01; First posted 2024-03-04 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: COVID-19
Keywords: CIC (Coronavirus Disease 2019 Influenza Combination); Influenza; Fluzone High-Dose
MeSH Terms: conditions — COVID-19; Influenza, Human | interventions — NVX-CoV2373 adjuvated lipid nanoparticle; Fluzone High-Dose; Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- CIC Vaccine (Experimental): A single 0.5 mL IM injection on Day 0
  Interventions: Biological: CIC Vaccine Co-formulated tNIV2 , SARSCoV-2 rS and Matrix-M Adjuvant
- Novavax COVID-19 Vaccine (Experimental): A single 0.5 mL IM injection on Day 0
  Interventions: Biological: Novavax COVID-19 Vaccine
- tNIV Vaccine (Experimental): A single 0.5 mL IM injection on Day 0
  Interventions: Biological: tNIV Vaccine
- Fluzone High-Dose (Experimental): A single 0.5 mL IM injection on Day 0
  Interventions: Biological: Fluzone High Dose

INTERVENTIONS:
Biological: CIC Vaccine Co-formulated tNIV2 , SARSCoV-2 rS and Matrix-M Adjuvant — CIC will contain SARs-CoV-2 antigen (35 μg), tNIV antigens (2 influenza A [H1N1 and H3N2] and 1 influenza B-Victoria lineage strains; 60 μg/strain
  Other Names: COVID-19 and influenza combination
  Arms: CIC Vaccine
Biological: Novavax COVID-19 Vaccine — Each 0.5 mL dose comprises 5 µg SARS-CoV-2 S protein and 50 µg Matrix-M adjuvant
  Other Names: Novavax SARS-CoV-2 rS vaccine
  Arms: Novavax COVID-19 Vaccine
Biological: tNIV Vaccine — 2 influenza A [H1N1 and H3N2] and 1 influenza B-Victoria lineage strains (60 μg/strain), and Matrix-M adjuvant (75 μg)
  Other Names: Trivalent Nanoparticle Influenza Hemagglutinin Vaccine
  Arms: tNIV Vaccine
Biological: Fluzone High Dose — Fluzone High-Dose is supplied as a suspension for IM injection 0.5 mL with 60 µg per strain
  Other Names: Fluzone HD
  Arms: Fluzone High-Dose

SUMMARY:
This is a medical study where participants will be randomly assigned to receive either a new combination vaccine that protects against both COVID-19 and the flu, or a standard flu vaccine. The researchers conducting the study won't know which vaccine each participant receives, ensuring their observations are unbiased. This study compares the new combination vaccine to an already available flu vaccine to see how well it works. It's a large-scale, final-stage study designed to thoroughly check how well the vaccines trigger an immune response (immunogenicity) and how safe they are.

DETAILED DESCRIPTION:
The study will enroll up to approximately 7,022,000 medically stable (based on history and physical examination) adult male and female participants ≥ 65 65 years of age in Part 1 and up to approximately 2,300 medically stable (based on history and physical examination) adult male and female participants ≥ 65 years of age in Part 2. In Part 1, pParticipants will be randomly assigned to receive either CIC, Novavax COVID-19 Vaccine, tNIV, or Fluzone High-Dose in a 3:2:1:3 ratio, respectively. All participants will receive a single intramuscular (IM) injection on Day 0, will remain on study for immunogenicity data collection through Day 182 and safety data collection through Day 364 (End of Study [EoS]).

ELIGIBILITY:
Inclusion Criteria

To be included in this study, each individual must satisfy all the following criteria:

1. Willing and able to give informed consent prior to study enrollment.
2. Medically stable adult male or female ≥ 65 years of age at Screening.
3. Participants may have 1 or more chronic medical diagnoses, but should be clinically stable as assessed by:

   1. Absence of changes in medical therapy in the past 2 months due to treatment failure or toxicity;
   2. Absence of medical events qualifying as SAEs within 3 months; and
   3. Absence of known, current, and life-limiting diagnoses which render survival to completion of the protocol unlikely in the opinion of the Investigator.
4. The participant has a body mass index (BMI) of 17 to 40 kg/m2, inclusive, at Screening.
5. Participant must be able to receive an injection in the deltoid of at least 1 arm.
6. Able to attend study visits, comply with study requirements, and provide reliable and complete reports of AEs.
7. Participants must have completed a primary vaccination series/booster against SARS CoV-2 with an authorized/approved COVID-19 vaccine, with receipt of last dose of authorized/approved vaccine (with or without boosters[s]) ≥ 8 weeks prior to vaccination.
8. Female participants must be surgically sterile (ie, have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or postmenopausal (defined as amenorrhea at least 12 consecutive months)
9. Participants must agree to not participate in any other SARS-CoV-2 or influenza prevention or treatment studies for the duration of the study. Note: For participants who become hospitalized with COVID-19 or influenza, participation in investigational treatment studies is permitted.

Exclusion Criteria

If an individual meets any of the following criteria, he or she is ineligible for this study:

1. History of laboratory-confirmed (by polymerase chain reaction [PCR], rapid antigen test, or rapid molecular assay) COVID-19, asymptomatic SARS-CoV-2 infection, or influenza within ≤ 8 weeks prior to Screening.
2. Any ongoing, symptomatic acute illness requiring medical or surgical care or chronic illness that required substantive changes in medication in the past 2 months prior to Screening indicating that chronic illness/disease is not stable (at the discretion of the investigator). This includes any current workup of undiagnosed illness that could lead to a new condition.
3. Serious chronic diseases inclusive of:

   1. Uncontrolled hypertension (NOTE: hypertension ≤ 170/100 is NOT exclusionary);
   2. Congestive heart failure requiring hospitalization within 3 months prior to Screening
   3. Chronic obstructive pulmonary disease (COPD) requiring hospitalization within 3 months prior to Screening (NOTE: stable COPD is NOT exclusionary);
   4. Within 3 months prior to Screening, evidence of unstable coronary artery disease as manifested by cardiac interventions (eg, cardiac stent placement, coronary artery bypass graft surgery), new cardiac medications for control of symptoms, or unstable angina (NOTE: stable coronary heart disease is NOT exclusionary);
   5. Hospitalization for diabetic ketoacidosis within 6 months prior to Screening
   6. Chronic kidney disease/renal requiring institution of substantive new therapy within 3 months prior to Screening
   7. Chronic clinically significant gastrointestinal and hepatic diseases requiring hospitalization or institution of substantive new therapy within 3 months prior to Screening. (for example, gastroesophageal reflux disease is NOT exclusionary)
   8. Chronic neurological diseases or neurological compromise preventing access to the study clinic, compliance with protocol, or accurate reporting of safety.
4. Participation in research involving an investigational product (drug/biologic/device) within 90 days before planned date of vaccination.
5. Use of COVID-19 prophylactic or treatment monoclonal antibodies or antibody cocktails within 90 days prior to planned date of vaccination.
6. History of a serious reaction to a prior influenza vaccination or known allergy to constituents of influenza vaccines - including egg proteins - or polysorbate 80; or any known allergies to products contained in the investigational product.
7. Any history of anaphylaxis to any prior vaccine.
8. History of Guillain-Barré Syndrome following a previous influenza vaccine.
9. Receipt of any vaccine in the 4 weeks preceding the study vaccination and any influenza vaccine within 2 months preceding the study vaccination. Note: Routine vaccinations will not be allowed until after study Day 21 and COVID-19 and influenza vaccination will not be allowed until after Day 84.
10. Any known or suspected autoimmune or immunosuppressive illness, congenital or acquired, based on medical history and/or physical examination (NOTE: well-controlled hypothyroidism and mild psoriasis are not exclusionary).
11. Chronic administration (defined as more than 14 continuous days) of immunosuppressants or other immune-modifying drugs within 6 months prior to the administration of the study vaccines. An immunosuppressant dose of glucocorticoid is defined as a systemic dose ≥ 10 mg of prednisone per day or equivalent. The use of topical, inhaled, and nasal glucocorticoids is permitted.
12. Administration of immunoglobulins and/or any blood products within the 3 months preceding the administration of the study vaccine or during the study.
13. Active cancer (malignancy) therapy within 1 year prior to study vaccination (with the exception of adequately treated non-melanomatous skin carcinoma or lentigo maligna and uterine cervical carcinoma in situ without evidence of disease, at the discretion of the investigator).
14. Participants who are breastfeeding, pregnant, or who plan to become pregnant prior to the EoS.
15. Suspected or known history of alcohol abuse or drug addiction within 2 years prior to study vaccination, which in the opinion of the investigator, might interfere with protocol compliance.
16. Acute disease at the time of enrollment (defined as the presence of a moderate or severe illness with or without fever, or an oral temperature ≥ 38.0°C, on the planned day of vaccine administration).
17. History of myocarditis or pericarditis.
18. Any condition that in the opinion of the investigator would pose a health risk to the participant if enrolled or could interfere with evaluation of the vaccine or interpretation of study results (including neurologic or psychiatric conditions deemed likely to impair the quality of safety reporting).
19. Study team member or immediate family member of any study team member (inclusive of Sponsor, Contract Research Organization, and study site personnel involved in the conduct or planning of the study).
20. Known history of any prior motor neuropathy.

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 9320 (Actual)
Dates: Start 2024-12-09 (Actual); Primary Completion 2026-07-26 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Numbers of participants with solicited local and systemic adverse events (AEs) | 7 days post-vaccination
  Numbers of participants with solicited local and systemic AEs over the 7 days post-vaccination.
Numbers of participants reporting unsolicited AEs and medically attended adverse events (MAAEs). | 28 days post-vaccination
  Numbers of participants reporting unsolicited AEs and MAAEs over 21 days post-vaccination.
Treatment-related MAAEs, serious adverse events (SAEs), and adverse events of special interest (AESIs) (including potential immune-mediated medical conditions [PIMMCs] and myocarditis and/or pericarditis) | Day 0 to Day 364
  Numbers of participants with treatment-related MAAEs, AESIs (including PIMMC and myocarditis and/or pericarditis), and SAEs will be collected for 12 months (approximately 364 days) post-vaccination.
Hemagglutination Inhibition (HAI) antibody responses of the CIC vaccine compared to Fluzone High-Dose of homologous A and B strains Expressed as GMT | Days 0 and 28
  Hemagglutination Inhibition (HAI) antibody responses of the CIC vaccine compared to Fluzone High-Dose of homologous influenza strains (two influenza A strains and one influenza B-Victoria lineage strain) on Days 0 and 28
Hemagglutination Inhibition (HAI) antibody responses of the CIC vaccine compared to Fluzone High-Dose of homologous A and B strains Expressed as GMTR | Days 28
  Hemagglutination Inhibition (HAI) antibody responses of the CIC vaccine compared to Fluzone High-Dose of homologous influenza strains (two influenza A strains and one influenza B-Victoria lineage strain) on Days 28
Percentage of Participants With a (HAI) antibody responses of the CIC vaccine compared to Fluzone High-Dose for 3 vaccine-homologous influenza strains Expressed as SCR | Days 28
  Percentage of Participants With a (HAI) antibody responses of the CIC vaccine compared to Fluzone High-Dose for 3 vaccine-homologous influenza strain on Days 28
Neutralizing Antibody (NAb) Responses of the CIC vaccine compared to Fluzone High-Dose of homologous A and B strains Expressed as GMT | Days 28
  Neutralizing Antibody (NAb) Responses Assessed against three homologous influenza strains (two influenza A strains and one influenza B-Victoria lineage strain) on Day 28
Neutralizing Antibody (NAb) Responses of the CIC vaccine compared to Fluzone High-Dose of homologous A and B strains Expressed as GMTR | Days 28
  Neutralizing Antibody (NAb) Responses Assessed against three homologous influenza strains (two influenza A strains and one influenza B-Victoria lineage strain) on Day 28
Percentage of Participants With a (NAb) Responses of the CIC vaccine compared to Fluzone High-Dose of homologous A and B strains Expressed as SCR | Days 28
  Neutralizing Antibody (NAb) Responses Assessed against three homologous influenza strains (two influenza A strains and one influenza B-Victoria lineage strain) on Day 28
Hemagglutination Inhibition (HAI) antibody titers specific to HA receptor-binding domains of (tNIV) comparable to Fluzone High-Dose of homologous influenza A and B strains expressed as GMT | Day 28
  Hemagglutination Inhibition (HAI) antibody titers specific to HA receptor-binding domains of (tNIV) comparable to Fluzone High-Dose of 2 influenza A strains and an influenza B-Victoria lineage strain) on Day 28
Hemagglutination Inhibition (HAI) antibody titers specific to HA receptor-binding domains of (tNIV) comparable to Fluzone High-Dose of homologous influenza A and B strains expressed as GMTR | Day 28
  Hemagglutination Inhibition (HAI) antibody titers specific to HA receptor-binding domains of (tNIV) comparable to Fluzone High-Dose of 2 influenza A strains and an influenza B-Victoria lineage strain) on Day 28
Percentage of Participants with (HAI) antibody titers specific to HA receptor-binding domains of (tNIV) comparable to Fluzone High-Dose of homologous influenza A and B strains expressed as SCR | Day 28
  Hemagglutination Inhibition (HAI) antibody titers specific to HA receptor-binding domains of (tNIV) comparable to Fluzone High-Dose of 2 influenza A strains and an influenza B-Victoria lineage strain) on Day 28

SECONDARY OUTCOMES:
Immunogenicity- HAI antibody titers specific for the HA receptor binding domains of vaccine homologous A and B influenza strains Expressed as Geometric Mean Titers (GMT) | Days 28
  HAI antibody titers specific for the HA receptor binding domains of vaccine response CIC vaccine compared to Fluzone High-Dose on Day 28
Immunogenicity- HAI antibody titers specific for the HA receptor binding domains of vaccine homologous A and B influenza strains Expressed as GMFR | Days 28
  HAI antibody titers specific for the HA receptor binding domains of vaccine response CIC vaccine compared to Fluzone High-Dose on Day 28
Percentage of Participants with HAI antibody titers specific for the HA receptor binding domains of vaccine homologous A and B influenza strains Expressed as SCR | Days 28
  HAI antibody titers specific for the HA receptor binding domains of vaccine response CIC vaccine compared to Fluzone High-Dose on Day 28
HAI antibody titers specific for the HA receptor binding domains of vaccine homologous A and B influenza strains Expressed as GMTR | Days 28
  HAI antibody titers specific for the HA receptor binding domains of vaccine response CIC vaccine compared to Fluzone High-Dose on Day 28
Influenza NAb responses: neutralizing antibody titers specific to vaccine homologous wild-type A and B influenza strains, is expressed as GMT | Days 28
  Neutralizing antibody titers specific to vaccine homologous influenza strains (ie, 2 influenza A strains and an influenza B-Victoria lineage strain) as measured by a neutralization assay, CIC and Fluzone High Dose on Day 28
Influenza NAb responses: neutralizing antibody titers specific to vaccine homologous wild-type A and B influenza strains, is expressed as GMFR | Days 28
  Neutralizing antibody titers specific to vaccine homologous influenza strains (ie, 2 influenza A strains and an influenza B-Victoria lineage strain) as measured by a neutralization assay, CIC and Fluzone High Dose on Day 28
Percentage of Participants with a NAb responses: neutralizing antibody titers specific to vaccine homologous wild-type A and B influenza strains, is expressed as SCR | Days 28
  Neutralizing antibody titers specific to vaccine homologous influenza strains (ie, 2 influenza A strains and an influenza B-Victoria lineage strain) as measured by a neutralization assay, CIC and Fluzone High Dose on Day 28
Influenza NAb responses: neutralizing antibody titers specific to vaccine homologous wild-type A and B influenza strains, is expressed as GMTR | Days 28
  Neutralizing antibody titers specific to vaccine homologous influenza strains (ie, 2 influenza A strains and an influenza B-Victoria lineage strain) as measured by a neutralization assay, CIC and Fluzone High Dose on Day 28
Hemagglutination Inhibition (HAI) antibody titers to tNIV and Fluzone High-Dose Expressed as GMT | Day 28
  Hemagglutination Inhibition (HAI) antibody titers specific to HA receptor-binding domains of vaccine-homologous influenza A and B strains on Day 28
Hemagglutination Inhibition (HAI) antibody titers to tNIV and Fluzone High-Dose Expressed as GMFR | Day 28
  Hemagglutination Inhibition (HAI) antibody titers specific to HA receptor-binding domains of vaccine-homologous influenza A and B strains on Day 28 homologous SARS-CoV-2 strain CIC, Fluarix or Fluzone HD, and Novavax COVID-19 Vaccine expressed as SCR
Percentage of Participants with (HAI) antibody titers to tNIV and Fluzone High-Dose Expressed as SCR | Day 28
  Hemagglutination Inhibition (HAI) antibody titers specific to HA receptor-binding domains of vaccine-homologous influenza A and B strains on Day 28
Influenza neutralizing antibody (NAb) responses of trivalent nanoparticle influenza vaccine (tNIV) comparable to Fluzone High-Dose Expressed as GMT | Day 28
  Influenza neutralizing antibody (NAb) responses of trivalent nanoparticle influenza vaccine (tNIV) comparable to Fluzone High-Dose against three influenza strains (two A strains and one B-Victoria strain) on Day 28.
Influenza neutralizing antibody (NAb) responses of trivalent nanoparticle influenza vaccine (tNIV) comparable to Fluzone High-Dose Expressed as GMFR | Day 28
  Influenza neutralizing antibody (NAb) responses of trivalent nanoparticle influenza vaccine (tNIV) comparable to Fluzone High-Dose against three influenza strains (two A strains and one B-Victoria strain) on Day 28.
Influenza neutralizing antibody (NAb) responses of trivalent nanoparticle influenza vaccine (tNIV) comparable to Fluzone High-Dose Expressed as GMTR | Day 28
  Influenza neutralizing antibody (NAb) responses of trivalent nanoparticle influenza vaccine (tNIV) comparable to Fluzone High-Dose against three influenza strains (two A strains and one B-Victoria strain) on Day 28.
Percentage of Participants with (NAb) responses of trivalent nanoparticle influenza vaccine (tNIV) comparable to Fluzone High-Dose Expressed as SCR | Day 28
  Influenza neutralizing antibody (NAb) responses of trivalent nanoparticle influenza vaccine (tNIV) comparable to Fluzone High-Dose against three influenza strains (two A strains and one B-Victoria strain) on Day 28.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development, Study Director — Novavax, Inc.
Locations (58):
- Australia (39):
  - Paratus Clinical Research - Canberra - PPDS, Bruce, Australian Capital Territory
  - Momentum Wellers, Wellers Hill, Brisbane
  - Paratus Clinical Research - Western Sydney - PPDS, Blacktown, New South Wales
  - Key Health- Bondi Junction, Bondi Junction, New South Wales
  - Emeritus Research - Sydney - PPDS, Botany, New South Wales
  - Genesis Research Services, Broadmeadow, New South Wales
  - Northern Beaches Clinical Research - PPDS, Brookvale, New South Wales
  - Northside Health, Coffs Harbour, New South Wales
  - East Sydney Doctors, Darlinghurst, New South Wales
  - Momentum Darlinghurst, Darlinghurst, New South Wales
  - Oztrials Clinical Research, Drummoyne, New South Wales
  - Paratus Clinical Research - Central Coast - PPDS, Kanwal, New South Wales
  - Novatrials, Kotara, New South Wales
  - Australian Clinical Research Network, Maroubra, New South Wales
  - Hunter Diabetes Centre, Merewether, New South Wales
  - Sutherland Shire Clinical Research - PPDS, Miranda, New South Wales
  - Pioneer Clinical Research - North Sydney, North Sydney, New South Wales
  - Taylor Square Private Clinic, Surry Hills, New South Wales
  - Momentum St Leonards, Sydney, New South Wales
  - Innovate Clinical Research Pty Ltd, Sydney, New South Wales
  - Wollongong Clinical Research - PPDS, Wollongong, New South Wales
  - Menzies School of Health Research, Casuarina, Northern Territory
  - University of the Sunshine Coast, Vitality Village - UniSC Clinical Trials - PPDS, Birtinya, Queensland
  - Momentum Taringa, Brisbane, Queensland
  - Griffith University Clinical Trials Unit, Griffith, Queensland
  - Nucleus Network Pty Ltd, Herston, Queensland
  - Paratus Clinical Research - Brisbane Clinic - PPDS, Herston, Queensland
  - Mater Hospital Brisbane, South Brisbane, Queensland
  - Cmax - Ppds, Adelaide, South Australia
  - Veritus Research - Emeritus - PPDS, Bayswater, Victoria
  - Emeritus Research -PPDS, Camberwell, Victoria
  - Ryrie St, Geelong, VIC 3220, Australia, Geelong, Victoria
  - Doherty Clinical Trials Limited, Melbourne, Victoria
  - Nucleus Network Limited, Melbourne, Victoria
  - Momentum Sunshine, Melbourne, Victoria
  - University of Melbourne - Melbourne, Melbourne N., Victoria
  - Institute for Respiratory Health - Midland, Midland, Western Australia
  - Telethon Kids Institute, Nedlands, Western Australia
  - CliniTrials, Perth, Western Australia
- New Zealand (19):
  - Momentum Tauranga - PPDS, Tauranga, Bay of Plenty
  - Momentum Hawke's Bay - PPDS, Hastings, Hawke's Bay Region
  - Momentum Dunedin - PPDS, Dunedin, Otago
  - Southern Clinical Trials - Totara - PCRN - PPDS, Auckland
  - Pacific Clinical Research Network - Auckland - PCRN - PPDS, Auckland
  - Optimal Clinical Trials Ltd - North Shore - PPDS, Auckland
  - Optimal Clinical Trials Ltd - PPDS, Auckland
  - Momentum Pukekohe - PPDS, Auckland
  - New Zealand Clinical Research - Christchurch - PPDS, Christchurch
  - Pacific Clinical Research Network - Christchurch - PCRN - PPDS, Christchurch
  - Lakeland Clinical Trials - Waikato - PCRN-PPDS, Hamilton
  - Momentum Lower Hutt - PPDS, Lower Hutt
  - Southern Clinical Trials - Tasman - PCRN - PPDS, Nelson
  - Momentum Palmerston North - PPDS, Palmerston North
  - Pacific Clinic Research Network - Rotorua - PCRN - PPDS, Rotorua
  - Momentum Kapiti - PPDS, Waikanae
  - Lakeland Clinical Trials - Wellington - PCRN - PPDS, Wellington
  - Momentum Wellington - PPDS, Wellington
  - Aotearoa Clinical Trials Trust, Wellington